CLINICAL TRIAL: NCT02031224
Title: Effect of Very Low Protein Diet Supplemented With Ketoanalogues of the Essential Amino Acids on the Progression of Chronic Kidney Disease
Brief Title: Supplemented Very Low Protein Diet and the Progression of Chronic Kidney Disease
Acronym: KETOPROG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Anemia Working Group Romania (Other)
Collaborators: Dr Carol Davila Teaching Hospital of Nephrology Bucharest (Unknown)
Responsible Party: Principal Investigator, Liliana Garneata, Assistant Professor of Nephrology, MD, PhD, Carol Davila University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AWG13/2007
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Restricted protein diets; Nutritional status
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — ketosteril; Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Keto-diet (KD) (Experimental): Patients in the intervention arm (KD group) will receive a vegetarian very low protein diet (0.3 g proteins/kg ideal body weight per day) supplemented with ketoanalogues of essential amino acids (Ketosteril®, Fresenius Kabi, Bad Homburg, Germany), 1 capsule for every 5 kg of ideal dry body weight per day.
  Interventions: Dietary Supplement: Very low protein diet supplemented with Ketosteril
- Low Protein Diet group (LPD) (Active Comparator): The patients in the control arm (LPD group) will continue their conventional low protein diet, with 0.6 g/kg per day (including high biological value proteins).
  The total recommended energy intake is of 30 kcal/kg of ideal dry body weight per day in both arms.
  Interventions: Behavioral: Conventional low protein diet

INTERVENTIONS:
Behavioral: Conventional low protein diet
  Other Names: LPD; Hypoproteic diet
  Arms: Low Protein Diet group (LPD)
Dietary Supplement: Very low protein diet supplemented with Ketosteril
  Other Names: SVLPD, Keto-diet
  Arms: Keto-diet (KD)

SUMMARY:
This is a prospective single center randomized controlled trial with a total duration of 18 months aiming to evaluate the effectiveness and the safety of a very low protein diet supplemented with ketoanalogues of essential aminoacids in reducing the progression of chronic kidney disease (CKD) in patients with advanced CKD.

DETAILED DESCRIPTION:
All eligible patients who will give informed consent will be screened. Those meeting the selection criteria will be enrolled and will enter a 3-month run-in phase during which a conventional LPD will be prescribed in all patients.

At the end of this phase, the subjects still fulfilling all the selection criteria will be randomized in a 1:1 ratio to receive the KD or to continue the conventional LPD for a total duration of 15 months.

Nineteen blood and urine samplings are scheduled for each patient, to be drawn monthly. The laboratory reports include the nitrogen compounds, calcium-phosphorus metabolism parameters, acid-base balance, biochemical nutritional markers, serum C-reactive protein, hemoglobin, blood cell count, and biochemical safety parameters (sodium, potassium, liver enzymes, and bilirubin).

The anthropometric measurements and subjective global assessment will be evaluated at enrolment, at randomization, and every 3 months thereafter.

The compliance with the prescribed diet (protein and energy intake) will be assessed monthly during the run-in phase, weekly for the first month after randomization, every 4 weeks during the next 6 months, and every 3 months thereafter.

The blood pressure levels, drugs required for the therapy of hypertension, acidosis and mineral metabolism disorders, and occurrence of adverse events will be recorded monthly.

ELIGIBILITY:
Inclusion Criteria:

* adult non-diabetic patients
* stage 4-5 CKD not on dialysis (estimated glomerular filtration by Modification of Diet in Renal Disease formula < 30 mL/min per year
* stable renal function at least 12 weeks before enrollment
* well-controlled arterial blood pressure
* proteinuria less than 1 g/g urinary creatinine
* good nutritional status
* declared and anticipated good compliance with the prescribed diet

Exclusion Criteria:

* poorly controlled arterial blood pressure (≥145/85 mm Hg)
* relevant comorbid conditions (diabetes mellitus, heart failure, active hepatic disease, digestive diseases with malabsorption, inflammation/anti-inflammatory therapy)
* uremic complications (pericarditis, polyneuropathy)
* feeding inability (anorexia, nausea)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2008-03; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Primary composite endpoint | 15 months after randomization
  Need for renal replacement therapy or an at least 50% reduction in the estimated glomerular filtration rate compared to randomization

SECONDARY OUTCOMES:
Secondary efficacy parameter | months 3-15 after randomization
  The rate of decline in the estimated Glomerular Filtration Rate
Secondary outcome measure - nitrogen balance | 15 months after randomization
  variations in serum urea
Secondary efficacy parameter - mineral metabolism | 15 weeks after randomization
  variations in total serum calcium
Secondary efficacy parameter | 15 weeks after randomization
  variations in serum phosphate level
Secondary efficacy parameter | 15 weeks after randomization
  variations in serum bicarbonate
Secondary safety parameter | 18 weeks after enrolment
  Subjective Global Assessment of the nutritional status
Secondary safety parameter | 18 weeks after enrolment
  Body Mass Index
Secondary outcome measure - Nutritional status | 18 weeks after enrolment
  Tricipital skinfold
Secondary safety parameter - anthropometric measures | 18 weeks after enrolment
  Mid-arm muscular circumference
Nutritional status - biochemical markers | 18 weeks after enrolment
  serum albumin
Inflammation | 18 weeks after enrolment
  serum level of C reactive protein
Nutritional status - biochemical marker | 18 weeks after enrolment
  Serum total cholesterol
Secondary safety parameter | 18 weeks after enrolment
  Serum potassium level
Secondary safety parameter | 18 weeks after enrolment
  liver enzymes: Aspartate Aminotransferase, Alanine Transaminase
Safety parameter - adverse events | 18 weeks after enrolment
  Occurrence of any adverse event
Secondary safety parameter - withdrawals | 18 weeks after enrolment
  number of withdrawals

OTHER OUTCOMES:
Compliance - protein intake | 18 months after enrolment
  urinary urea nitrogen excretion to calculate the protein intake
Compliance - energy intake | 18 weeks after enrolment
  3-day food diary to calculate the daily energy intake

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Mircescu, Prof, Study Chair — Carol Davila University of Medicine and Pharmacy
Locations (1):
- "Dr Carol Davila" Teaching Hospital of Nephrology, Bucharest, Romania

REFERENCES:
- [Result] Mircescu G, Garneata L, Stancu SH, Capusa C. Effects of a supplemented hypoproteic diet in chronic kidney disease. J Ren Nutr. 2007 May;17(3):179-88. doi: 10.1053/j.jrn.2006.12.012. PMID 17462550
- [Derived] Hahn D, Hodson EM, Fouque D. Low protein diets for non-diabetic adults with chronic kidney disease. Cochrane Database Syst Rev. 2020 Oct 29;10(10):CD001892. doi: 10.1002/14651858.CD001892.pub5. PMID 33118160